CLINICAL TRIAL: NCT02239055
Title: Staff Nurse Perceptions of the Impact of Mentalization Based Treatment (MBT) Skills Training on Clinical Practice When Working With Borderline Personality Disorder (BPD) in Acute Mental Health Admission Wards: A Qualitative Analysis.
Brief Title: Staff Nurse Perceptions of MBT Skills Training for Working With BPD in AMH
Status: Completed | Type: Observational
Sponsor: University of Aberdeen (Other)
Collaborators: NHS Grampian (Other Government)
Responsible Party: Sponsor
Other Study IDs: 14/NS/0063
Record Dates: First submitted 2014-09-08; First posted 2014-09-12 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2014-09

CONDITIONS: Borderline Personality Disorder
Keywords: Borderline Personality Disorder; Mentalization Based Treatment; MBT Skills Training; Staff Nurse Perceptions; Acute Mental Health
MeSH Terms: conditions — Borderline Personality Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Focus Group 1: Staff Perceptions
- Focus Group 2: Staff Perceptions

SUMMARY:
Despite expert opinion unconvinced of any value for hospitalization in caring for people with borderline personality disorder (BPD), this patient group still accounts for a significant proportion of adult acute mental health (AMH) admissions. Staff nurses generally voice negative perceptions of BPD, a view which is linked to an uncertainty of how to approach these patients, and difficulties leading to personal distress and burnout. Mentalization-based treatment (MBT) is an evidence based approach, focusing on the mental states of both self and others, developed specifically to treat BPD and facilitated successfully in specialised settings. MBT Skills training is a compact and cost effective two day workshop which equips generalist mental health nurses with a skillset enabling them to work effectively with BPD. MBT Skills training was first offered to staff nurses in Royal Cornhill Hospital, Aberdeen in 2013. This study aims to assess staff perceptions on the value of MBT skills training, evaluating how it impacts on clinical practice when working with BPD in AMH.

DETAILED DESCRIPTION:
Methodology: Using two focus groups with a neutral facilitator, a purposive sample of nine staff nurses took part in a semi-structured exploration of BPD in AMH. Participants discussed challenges with patients and the impact of MBT skills training and Clinical Supervision (CS). The focus groups were audio recorded and transcribed verbatim. Data was examined using a thematic analysis.

ELIGIBILITY:
Inclusion Criteria:

* Staff nurses aged between 18 and 65, who had completed the 2 day Mentalization Based Treatment (MBT) skills training and were still working in acute mental health.

Exclusion Criteria:

* Staff nurses under 18 or over 65, who had not completed the 2 day Mentalization Based Treatment (MBT) skills training and were not working in acute mental health.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Staff nurses who had completed the 2 day Mentalization Based Treatment (MBT) skills training and were still working in acute mental health.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2014-05; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Focus Groups | 2 hours for focus groups, one month data analysis
  Focus Groups used to measure Staff nurse perceptions of the impact of MBT and associated issues in working with BPD in AMH.

CONTACTS AND LOCATIONS:
Overall Officials: Dan Warrender, BN, MA, Principal Investigator — NHS Grampian / University of Aberdeen
Locations (1):
- Royal Cornhill Hospital, Aberdeen, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided